CLINICAL TRIAL: NCT02961660
Title: An Open-label Study to Evaluate the Effect of Severe Renal Impairment on the Single-dose Pharmacokinetics of Odalasvir
Brief Title: A Study to Evaluate the Effect of Severe Renal Impairment on the Single-dose Pharmacokinetics of Odalasvir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108242; 64294178HPC1014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — odalasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Severe Renal Impairment): Odalasvir (Experimental): Participants will receive single oral dose of odalasvir 25 milligram (mg) under fed conditions (standard breakfast) on Day 1.
  Interventions: Drug: Odalasvir
- Cohort 2 (Normal Renal Function): Odalasvir (Experimental): Participants will receive single oral dose of odalasvir 25 milligram (mg) under fed conditions (standard breakfast) on Day 1.
  Interventions: Drug: Odalasvir

INTERVENTIONS:
Drug: Odalasvir — Participants will receive odalasvir 25 mg tablet, orally.

SUMMARY:
The main purpose of this study is to evaluate the pharmacokinetics (PK) of a single oral dose of odalasvir (ODV) in participants with severe renal impairment and compare with the PK in matched participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

Cohorts 1 and 2:

* Participant must have a body mass index (BMI; weight in kilogram (kg) divided by the square of height in meters) of 18 to 36 kilogram per meter square (kg/m^2), extremes included, and a body weight not less than 50.0 kg
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in the protocol
* Male Participant must agree not to donate sperm from enrollment (Day 1) in the study until at least 30 days after receiving the study drug
* Female Participant, except if postmenopausal, must have a negative serum (beta human chorionic gonadotropin [beta hCG]) pregnancy test at screening and negative highly sensitive urine pregnancy test at Day -1

Cohort 1:

* Participant must have severe renal impairment not requiring dialysis, defined as an estimated glomerular filtration rate (eGFR) less than (<) 30 milliLiter per minute (mL/min)/1.73 m^2
* Participant must have stable renal function that is no significant change in renal function as evidenced by the (mean) screening serum creatinine value within +/-25 percent (%) from the determination obtained at least 3 months prior to screening, and expected to remain stable during the study, and not be planning to initiate dialysis during the study period
* Participant must be otherwise healthy except for renal impairment and its underlying disease states and mild comorbidities and participant must be medically stable on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening. If there are abnormalities or results outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

Cohort 2:

* Participant must be healthy on the basis of physical examination, medical history, vital signs, 12-lead ECG, and clinical laboratory tests performed at screening
* Participant must have an eGFR greater than or equal to (>=) 90 mL/min/1.73 m^2

Exclusion Criteria:

Cohorts 1 and 2:

* Participant has a history of any illness (unrelated to renal impairment or its underlying disease, as appropriate) that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant. This may include but is not limited to history of relevant drug or food allergies, history of cardiovascular or central nervous system disease, history or presence of clinically significant pathology, chronic skin disease, or history of mental disease
* Participant who is on a vegetarian diet or who takes creatine supplements, and who has a non-standard muscle mass, example amputation, malnutrition, muscle wasting, or extremely muscular (body building)
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening
* Participant has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening
* Participant who smokes more than 10 cigarettes or 2 cigars or 2 pipes per day from within 3 months before screening until the end of the study
* Participant is a woman who is pregnant, or breast-feeding, or planning to become pregnant from signing of the informed consent form (ICF) onwards until 30 days after study drug administration
* Participant is a man who plans to father a child while enrolled in this study (Day 1) until 30 days after study drug administration

Cohort 1:

* Participant requires dialysis
* Participant with imminent renal replacement therapy (that is, during the study period)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  The Cmax is the maximum observed plasma analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours.
Area Under the Plasma Concentration-Time Curve From Time Zero to 72 Hours (AUC[0-72]) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  The AUC (0-72) is the area under the plasma concentration-time curve from time zero to 72 hours.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Apparent Elimination Half-Life (t1/2) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  Elimination half-life associated with the terminal slope Lambda (z) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda (z).
Apparent Volume of Distribution (Vd/F) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Total Apparent Oral Clearance (CL/F) of Odalasvir | Predose and 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 60, 72, 96 120, 144, 168, and 312 hours postdose
  The CL/F is defined as Dose/AUC (0-infinity).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Baseline, up to follow-up (30 to 35 days after study drug intake)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Orlando, Florida
  - Knoxville, Tennessee